CLINICAL TRIAL: NCT01398059
Title: The Metabolic Effects of Breaks in Sedentary Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Mark Tremblay, Dr Mark Tremblay, Director, Healthy Active Living and Obesity Research Group, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11/01E
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-05

CONDITIONS: Feasibility; Insulin; Glucose; Lipids; Eating
Keywords: Sedentary Behavior; Cardiometabolic Risk; Pediatrics
MeSH Terms: conditions — Insulin Resistance; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sedentary (Experimental): In this condition, participants will engage in 8 hours of uninterrupted sedentary behaviour.
  Interventions: Other: Sedentary
- Sedentary With Breaks (Experimental): In this condition participants will engage in 8 hours of sitting, although the sitting will be interrupted every 20 minutes. During these interruptions participants will spend 2 minutes walking at an intensity equivalent to 30% of VO2peak.
  Interventions: Other: Sedentary With Breaks
- Sedentary With Breaks and Physical Activity (Experimental): In this condition participants will engage in 8 hours of sitting, although the sitting will be interrupted every 20 minutes. During these interruptions participants will spend 2 minutes walking at an intensity equivalent to 30% of VO2peak. Participants will also engage in 20 minutes of structured physical activity at an intensity of 60% of VO2peak in both the morning and afternoon.
  Interventions: Other: Sedentary With Breaks and Physical Activity

INTERVENTIONS:
Other: Sedentary — In this condition, participants will engage in 8 hours of uninterrupted sedentary behaviour.
  Arms: Sedentary
Other: Sedentary With Breaks — In this condition participants will engage in 8 hours of sitting, although the sitting will be interrupted every 20 minutes. During these interruptions participants will spend 2 minutes walking at an intensity equivalent to 30% of VO2peak.
  Arms: Sedentary With Breaks
Other: Sedentary With Breaks and Physical Activity — In this condition participants will engage in 8 hours of sitting, although the sitting will be interrupted every 20 minutes. During these interruptions participants will spend 2 minutes walking at an intensity equivalent to 30% of VO2peak. Participants will also engage in 20 minutes of structured physical activity at an intensity of 60% of VO2peak in both the morning and afternoon.
  Arms: Sedentary With Breaks and Physical Activity

SUMMARY:
The purpose of this study is to determine whether acute bouts of sedentary behaviour (with or without breaks and/or structured physical activity) result in measurable changes in metabolic health in children and youth.

DETAILED DESCRIPTION:
North American children spend the majority of their waking hours engaging in sedentary behavior (e.g. sitting). Research in adults and animal models suggests that even short bouts of uninterrupted siting may result in acute changes increases in cardiometabolic risk, although to date no studies have investigated this relationship in children and youth. The purpose of this study is to assess the feasibility of a protocol which will expose participants aged 10-14 years to a full day of uninterrupted sitting, and to determine the impact of this protocol on markers of cardiometabolic risk (insulin, glucose, triglyceride, HDL-C and LDL-C) as well as subsequent food intake and physical activity. The impact of uninterrupted sitting will be compared to the impact of interrupted sitting, with and without the inclusion of moderate physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-14
* Normal weight or obese

Exclusion Criteria:

* Overweight
* Overt diabetes or heart disease (or taking medications to treat this conditions)
* Being unambulatory or otherwise unable to perform the study protocol

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Tremblay, OhD, Principal Investigator — Children's Hospital of Eastern Ontario Research Institute
Locations (1):
- Behavioural Metabolic Research Unit, University of Ottawa, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Saunders TJ, Chaput JP, Goldfield GS, Colley RC, Kenny GP, Doucet E, Tremblay MS. Prolonged sitting and markers of cardiometabolic disease risk in children and youth: a randomized crossover study. Metabolism. 2013 Oct;62(10):1423-8. doi: 10.1016/j.metabol.2013.05.010. Epub 2013 Jun 15. PMID 23773981

RESULTS

PARTICIPANT FLOW:
Groups:
- Sed, Sed With Breaks, Sed With Breaks and PA: In this condition, participants experienced the experimental conditions in the following order. Each condition was separated by at least 1 week.
  Sedentary condition
  Sedentary with breaks condition
  Sedentary with breaks and physical activity condition
- Sed, Sed With Breaks and PA, Sed With Breaks: In this condition, participants experienced the experimental conditions in the following order. Each condition was separated by at least 1 week.
  Sedentary condition
  Sedentary with breaks and physical activity condition
  Sedentary with breaks condition
- Sed With Breaks, Sed With Breaks and PA, Sed; Sed With Breaks and PA, Sed With Breaks, Sed: In this condition, participants experienced the experimental conditions in the following order. Each condition was separated by at least 1 week.
  Sedentary with breaks and physical activity condition
  Sedentary with breaks condition
  Sedentary condition
- Sed With Breaks, Sed, Sed With Breaks and PA: In this condition, participants experienced the experimental conditions in the following order. Each condition was separated by at least 1 week.
  Sedentary with breaks condition
  Sedentary condition
  Sedentary with breaks and physical activity condition
- Sed With Breaks and PA, Sed, Sed With Breaks: In this condition, participants experienced the experimental conditions in the following order. Each condition was separated by at least 1 week.
  Sedentary with breaks and physical activity condition
  Sedentary condition
  Sedentary with breaks condition
Period: Overall Study
Arm/Group | Sed, Sed With Breaks, Sed With Breaks and PA | Sed, Sed With Breaks and PA, Sed With Breaks | Sed With Breaks, Sed With Breaks and PA, Sed | Sed With Breaks, Sed, Sed With Breaks and PA | Sed With Breaks and PA, Sed, Sed With Breaks | Sed With Breaks and PA, Sed With Breaks, Sed
Started | 4 | 3 | 4 | 2 | 4 | 2
Completed | 4 | 3 | 4 | 2 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants experienced all 3 conditions, in random order.
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 19
Body Mass Index calculated using height and weight [Mean (Standard Deviation); unit: kg/m^2] | 18 (4)
Waist circumference measured in cm [Mean (Standard Deviation); unit: Centimetres] | 64 (12)
Pubertal stage measured by self-reported Tanner stage [Mean (Standard Deviation); unit: units on a scale] — Tanner stages are a scale of physical development in children, adolescents and adults. The scale ranges from 1 (pre-pubescent child) to 5 (adult), and defines physical measurements of development based on external primary and secondary sex characteristics, such as the size of the breasts, genitals, testicular volume and development of pubic hair.
  units on a scale | 2 (1)
Baseline PA level by Actical Accelerometer [Mean (Standard Deviation); unit: minutes/day] | 64 (27)
Baseline Sedentary Behaviour by Actical Accelerometer [Mean (Standard Deviation); unit: minutes/day] | 507 (56)
Insulin [Mean (Standard Deviation); unit: pmol/L] | 39 (24)
Glucose [Mean (Standard Deviation); unit: pmol/L] | 5 (0)
LDL-Cholesterol [Mean (Standard Deviation); unit: pmol/L] | 2 (1)
HDL-Cholesterol [Mean (Standard Deviation); unit: pmol/L] | 1 (1)
Triglycerides [Mean (Standard Deviation); unit: pmol/L] | 1 (0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Net Incremental Area-Under-The-Curve (iAUC)
Description: Insulin levels will be assessed multiple times throughout the day, and the resulting values will be used to calculate AUC.
Time Frame: Baseline, 1.5, 3, 4.5, 6, and 7.5 hours
Measure: Mean (Standard Deviation); unit: pmol/L/min
Arm/Group | Sedentary | Sedentary With Breaks | Sedentary With Breaks and Physical Activity
Number analyzed (Participants) | 19 | 19 | 19
pmol/L/min | 80559.3 (66380.3) | 78707.3 (83074.5) | 64270.8 (42272.4)

2. Secondary Outcome: Change in Triglyceride Net Incremental Area-Under-The-Curve (iAUC)
Description: Blood draws will be taken several times throughout the day, and the resulting values will be used to calculate AUC.
Time Frame: Baseline, 1.5, 3, 4.5, 6, and 7.5 hours
Measure: Mean (Standard Deviation); unit: mmol/L/min
Arm/Group | Sedentary | Sedentary With Breaks | Sedentary With Breaks and Physical Activity
Number analyzed (Participants) | 19 | 19 | 19
mmol/L/min | 99.8 (114.4) | 101.5 (69.0) | 65.2 (66.4)

3. Secondary Outcome: Change in HDL-Cholesterol (HDL-C) Net Incremental Area-Under-The-Curve (iAUC)
Description: Blood draws will occur throughout the day, and the resulting values will be used to calculate AUC.
Time Frame: Baseline, 1.5, 3, 4.5, 6, and 7.5 hours
Measure: Mean (Standard Deviation); unit: mmol/L/min
Arm/Group | Sedentary | Sedentary With Breaks | Sedentary With Breaks and Physical Activity
Number analyzed (Participants) | 19 | 19 | 19
mmol/L/min | -38.7 (39.9) | -32.2 (40.2) | -52.3 (41.4)

4. Secondary Outcome: Change in LDL-Cholesterol (LDL-C) Net Incremental Area-Under-The-Curve (iAUC)
Description: Blood draws will occur throughout the day, and the resulting values will be used to calculate AUC.
Time Frame: Baseline, 1.5, 3, 4.5, 6, and 7.5 hours
Measure: Mean (Standard Deviation); unit: mmol/L/min
Arm/Group | Sedentary | Sedentary With Breaks | Sedentary With Breaks and Physical Activity
Number analyzed (Participants) | 19 | 19 | 19
mmol/L/min | -62.9 (67.2) | -50.0 (28.9) | -76.5 (51.4)

5. Secondary Outcome: Change in Glucose Net Incremental Area-Under-The-Curve (iAUC)
Description: Blood draws will occur throughout the day, and the resulting values will be used to calculate AUC.
Time Frame: Baseline, 1.5, 3, 4.5, 6, and 7.5 hours
Measure: Mean (Standard Deviation); unit: mmol/L/min
Arm/Group | Sedentary | Sedentary With Breaks | Sedentary With Breaks and Physical Activity
Number analyzed (Participants) | 19 | 19 | 19
mmol/L/min | 185.3 (171.7) | 163.2 (148.8) | 248.0 (220.4)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Sedentary | Sedentary With Breaks | Sedentary With Breaks and Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No